CLINICAL TRIAL: NCT01930942
Title: Genetic Profile on Predicting Sensibility of Preoperative Chemoradiotherapy on Locally Advanced Rectal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Vice Director of Abdomen Division, Radiation Oncology Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0905001040531
Record Dates: First submitted 2013-08-14; First posted 2013-08-29 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Rectal Neoplasms
Keywords: rectal carcinoma; preoperative concurrent chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- preoperative concurrent chemoradiation (Experimental): Radiation is given with 5000 cGy in 25 fractions (5 weeks). Concurrent chemotherapy consists of oxaliplatin (50 mg/m2 ) intravenously over 2 h on days 1, 8, 15, 22 and 29, and capecitabine (825 mg/m2 twice day) was given orally on each day of radiation.
  Interventions: Radiation: preoperative concurrent chemoradiation

INTERVENTIONS:
Radiation: preoperative concurrent chemoradiation — Radiation is given with 5000 cGy in 25 fractions (5 weeks). Concurrent chemotherapy consists of oxaliplatin (50 mg/m2 ) intravenously over 2 h on days 1, 8, 15, 22 and 29, and capecitabine (825 mg/m2 twice day) was given orally on each day of radiation.

SUMMARY:
The aim of this study is to find some genetic factors in predicting the sensibility of preoperative chemoradiotherapy for locally advanced rectal carcinoma.

DETAILED DESCRIPTION:
For locally advanced rectal carcinoma,preoperative chemoradiotherapy(CRT) achieved similar overall survival and better local control compared with postoperative therapy,so it was considered to be one of the standard therapy of these patients.But,not every one will be cured,the possible reason is the difference gene expression and mutation status among patients.So,we performed this trial to study the relationship between genetic factors and response of preoperative CRT for locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed rectal adenocarcinoma, preoperative stage II / III (T3-4N0 or T1-4N + M0).
* Distance from the lower bound of tumor to the anal verge is less than 12 cm.
* KPS score not less than 70
* Can be tolerated chemotherapy and radiotherapy.
* No history of radiation therapy to the pelvis.
* Non-allergic history of fluorouracil or platinum-based chemotherapy drugs.
* Full understanding of the study, the ability to complete all of the treatment plan, follow up the conditions and sign the informed consent. -

Exclusion Criteria:

* Other malignancy (past or at the same time), does not include curable non-melanoma skin cancer and cervical carcinoma in situ; does not include resectable primary colon cancer (synchronous or metachronous).
* Pregnant or lactating patients.
* Fertility but did not use contraceptive measures.
* Existing active infection.
* Merge serious complications, can not tolerate the treatment, such as 6 months of myocardial infarction, mental illness, uncontrollable diabetes or uncontrollable hypertension or hypotension.
* Concurrent treatment with other anticancer drugs.
* Can not complete treatment or follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
gene expression in different response groups | 6 months after radical surgery

SECONDARY OUTCOMES:
overall survival, disease free survival and local-regional free survival | 3 years after pre-operative chemoradiotherapy

OTHER OUTCOMES:
toxicity | during concurrent chemoradiation
  any G3/4 toxicities according to CTC 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China